CLINICAL TRIAL: NCT07258030
Title: Development of a Decision Algorithm for Vital Sign Assessment in the Outpatient Physical Therapy Setting: An e-Delphi Study
Brief Title: Decision Algorithm for Vital Sign Assessment in the Outpatient Physical Therapy Setting
Status: Recruiting | Type: Observational
Sponsor: Youngstown State University (Other)
Responsible Party: Principal Investigator, Edmund Ickert, Primary Investigator, Youngstown State University
Other Study IDs: 2026-90
Record Dates: First submitted 2025-11-18; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Healthy
Keywords: delphi; vital sign; assessment; algorithm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physical Therapists in an Outpatient Setting: Expert Panel Cohort:
  Participants will be licensed physical therapists who meet the following inclusion criteria:
  1. Minimum of 5 years of clinical experience in an outpatient physical therapy setting.
  2. Proficient in English (reading and writing).
  3. Willing to provide informed consent and complete all survey rounds.
  Interventions: Other: E-Delphi

INTERVENTIONS:
Other: E-Delphi — Description:
  Round 1: Participants provide open-ended responses identifying signs, symptoms, and factors influencing decisions to assess or not assess vital signs.
  Round 2: Participants rank the importance of these factors using a 5-point Likert scale and may suggest additional items.
  Round 3: Participants review aggregated results and finalize consensus on criteria for inclusion in a decision algorithm.
  Mode of Delivery: Online survey via Qualtrics. Duration: Each round will remain open for 3 weeks, with reminder emails sent during weeks 1 and 2.

SUMMARY:
Brief Summary The goal of this observational study is to develop consensus-based criteria for when vital sign assessment (VSA) should be performed in outpatient physical therapy settings. The primary purpose is to identify clinical signs, symptoms, and other factors that inform decision-making for VSA to improve patient safety and guide treatment progression.

Main Questions:

1. Which clinical characteristics indicate that vital signs should be assessed during outpatient physical therapy?
2. Which clinical characteristics indicate that vital signs do not need to be assessed?

Study Design:

This study uses a three-round electronic Delphi (e-Delphi) process to achieve expert consensus.

Comparison:

Researchers will compare responses across rounds to determine agreement and stability of criteria for inclusion in a decision algorithm.

Participants:

Licensed physical therapists with ≥5 years of clinical experience in outpatient settings.

Procedures:

Participants will:

Complete three rounds of online surveys via Qualtrics. Round 1: Suggest signs, symptoms, and factors for assessing or not assessing vitals.

Round 2: Rank importance of these factors on a 5-point Likert scale and suggest additional items.

Round 3: Review aggregated results and finalize consensus on criteria.

DETAILED DESCRIPTION:
Vital sign assessment (VSA) in outpatient physical therapy settings is underutilized despite its potential to improve patient safety and guide clinical decision-making. Physical therapists often rely on subjective patient reports rather than objective measures such as blood pressure, heart rate, and oxygen saturation. Evidence suggests that VSA can identify cardiovascular complications, detect early signs of physiological distress, and inform exercise intensity adjustments during treatment sessions. In the post-COVID-19 era, where direct access to physical therapy is common, integrating VSA into routine practice may help identify conditions such as postural orthostatic tachycardia syndrome, hypertension, and exertional desaturation that could otherwise go unnoticed.

Currently, there are no standardized criteria to guide outpatient physical therapists on when VSA is necessary. This study aims to fill that gap by developing a decision algorithm based on expert consensus. Using a three-round electronic Delphi (e-Delphi) process, the study will engage experienced outpatient physical therapists to identify and prioritize clinical signs, symptoms, and contextual factors that should influence VSA decisions.

Study Objectives:

1. Generate a comprehensive list of factors that indicate when vital signs should or should not be assessed.
2. Achieve expert consensus on which factors should be included in a decision-making algorithm for VSA.

Methods:

Participants will be licensed physical therapists with at least five years of outpatient clinical experience. Recruitment will occur nationally through professional networks, state associations, and social media. The e-Delphi process will be conducted via Qualtrics and will include three rounds:

Round 1: Participants suggest signs, symptoms, and factors influencing VSA decisions.

Round 2: Participants rank the importance of these factors on a 5-point Likert scale and may propose additional items.

Round 3: Participants review aggregated results and finalize consensus on criteria.

Consensus will be evaluated using descriptive and inferential statistics, including median, interquartile range, percent agreement, Kendall's coefficient of concordance, and stability measures across rounds. Statements achieving consensus will form the basis of a decision algorithm for VSA in outpatient physical therapy.

Significance:

This study will provide evidence-based guidance for outpatient physical therapists, promoting safer and more effective care by standardizing VSA practices. The resulting algorithm may improve early detection of physiological abnormalities, optimize treatment progression, and enhance patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Licensed physical therapist.
2. Minimum of 5 years of clinical experience in an outpatient physical therapy setting.
3. Proficient in English (reading and writing).
4. Ability to provide informed consent.

Exclusion Criteria:

1. Less than 5 years of outpatient physical therapy experience.
2. Inability to read or write in English.
3. Declines informed consent or does not agree to participate in all survey rounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of licensed physical therapists who are considered experts in outpatient care. To qualify, participants must have at least five years of clinical experience in an outpatient physical therapy setting, and be proficient in English for reading and writing. All participants must provide informed consent and agree to complete three rounds of the e-Delphi survey process.
  Recruitment will occur nationally through professional networks, including American Board of Physical Therapy Specialties (ABPTS) listservs, state physical therapy associations, licensure boards, and social media outreach. Snowball sampling will be used by encouraging participants to share the study invitation with other eligible colleagues. The target population represents experienced clinicians who can provide expert input on decision-making for vital sign assessment in outpatient physical therapy.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-21 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Consensus on Criteria for Vital Sign Assessment | Approximately 9 weeks after initiation of Round 1 (end of Round 3).
  Determine which clinical signs, symptoms, and contextual factors should be included in a decision algorithm for vital sign assessment in outpatient physical therapy.
  Metric: Consensus defined as:
  Median ≥ 4 (agreement) or ≤ 2 (disagreement) Interquartile Range (IQR) ≤ 1 Percent Agreement ≥ 75% in Round 2 and ≥ 80% in Round 3

SECONDARY OUTCOMES:
Level of Agreement Among Experts | Approximately 9 weeks after initiation of Round 1 (end of Round 3).
  Measure overall agreement across all items and categories. Metric: Kendall's Coefficient of Concordance (W), where 0 = no agreement and 1 = perfect agreement (p ≤ 0.05 for significance).
Stability of Responses Between Rounds | Approximately 9 weeks after initiation of Round 1 (end of Round 3).
  Assess consistency of expert ratings between Round 2 and Round 3 Metric: Wilcoxon rank-sum test (p ≤ 0.05) and Intraclass Correlation Coefficient (ICC).

CONTACTS AND LOCATIONS:
Locations (1):
- Youngstown State University, Youngstown, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shang Z. Use of Delphi in health sciences research: A narrative review. Medicine (Baltimore). 2023 Feb 17;102(7):e32829. doi: 10.1097/MD.0000000000032829. PMID 36800594
- [Background] Severin R, Sabbahi A, Albarrati A, Phillips SA, Arena S. Blood Pressure Screening by Outpatient Physical Therapists: A Call to Action and Clinical Recommendations. Phys Ther. 2020;100:1008-1019. Phys Ther. 2021 Jul 1;101(7):pzaa122. doi: 10.1093/ptj/pzaa122. No abstract available. PMID 34279665
- [Background] Serdar CC, Cihan M, Yucel D, Serdar MA. Sample size, power and effect size revisited: simplified and practical approaches in pre-clinical, clinical and laboratory studies. Biochem Med (Zagreb). 2021 Feb 15;31(1):010502. doi: 10.11613/BM.2021.010502. Epub 2020 Dec 15. PMID 33380887
- [Background] Niederberger M, Spranger J. Delphi Technique in Health Sciences: A Map. Front Public Health. 2020 Sep 22;8:457. doi: 10.3389/fpubh.2020.00457. eCollection 2020. PMID 33072683
- [Background] Nasa P, Jain R, Juneja D. Delphi methodology in healthcare research: How to decide its appropriateness. World J Methodol. 2021 Jul 20;11(4):116-129. doi: 10.5662/wjm.v11.i4.116. eCollection 2021 Jul 20. PMID 34322364
- [Background] Gallotti M, Campagnola B, Cocchieri A, Mourad F, Heick JD, Maselli F. Effectiveness and Consequences of Direct Access in Physiotherapy: A Systematic Review. J Clin Med. 2023 Sep 7;12(18):5832. doi: 10.3390/jcm12185832. PMID 37762773
- [Background] Faletra A, Bellin G, Dunning J, Fernandez-de-Las-Penas C, Pellicciari L, Brindisino F, Galeno E, Rossettini G, Maselli F, Severin R, Mourad F. Assessing cardiovascular parameters and risk factors in physical therapy practice: findings from a cross-sectional national survey and implication for clinical practice. BMC Musculoskelet Disord. 2022 Aug 4;23(1):749. doi: 10.1186/s12891-022-05696-w. PMID 35927658
- [Background] Severin R, Wang E, Wielechowski A, Phillips SA. Outpatient Physical Therapist Attitudes Toward and Behaviors in Cardiovascular Disease Screening: A National Survey. Phys Ther. 2019 Jul 1;99(7):833-848. doi: 10.1093/ptj/pzz042. PMID 30883642
- [Background] Albarrati AM PT, PhD. Outpatient physical therapy cardiovascular assessment: Physical therapist perspective and experience. Physiother Theory Pract. 2019 Sep;35(9):843-850. doi: 10.1080/09593985.2018.1458355. Epub 2018 Mar 29. PMID 29596007